CLINICAL TRIAL: NCT00668733
Title: Follow-up Study to Evaluate Sustained Clearance Rates of Actinic Keratoses up to One Year After Completion of Studies GW01-0702, GW01-0703, GW01-0704, and GW01-0705
Brief Title: Follow-up Study to Evaluate Sustained Clearance Rates of Actinic Keratoses up to One Year
Status: Completed | Type: Observational
Sponsor: Graceway Pharmaceuticals, LLC (Industry)
Responsible Party: Sharon Levy, MD / Vice President, Product Development, Graceway Pharmaceuticals, LLC
Other Study IDs: GW01-0803
Record Dates: First submitted 2008-04-24; First posted 2008-04-29 (Estimated); Results first posted 2010-07-13 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Actinic Keratoses
Keywords: Actinic keratoses; Dermatologic disease
MeSH Terms: conditions — Keratosis, Actinic; Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study was to obtain long-term sustained clearance rates for subjects previously treated with imiquimod creams in studies GW01-0702, GW01-0703, GW01-0704 and GW01-0705.

DETAILED DESCRIPTION:
This is a Phase 3 longitudinal and observational study. Subjects who previously enrolled in studies GW01-0702, GW01-0703, GW01-0704, and GW01-0705 and were completely cleared of their AK lesions in the selected treatment area at the end-of-study visit will return for follow-up visits at 6 and 12 months after the EOS visit or until a recurrence of AKs.

The NCT numbers for the above mentioned studies are:

NCT00603798 - for Studies GW01-0703 and GW01-0705

NCT00605176 for Studies GW01-0702 and GW01-0704

ELIGIBILITY:
Inclusion Criteria:

* Are willing and able to give informed consent;
* Have successfully completed one of the following studies: GW01-0702, GW01- 0703, GW01-0704, or GW01-0705 and have been determined to be completely clear of AK lesions at the EOS visit in the designated treatment area from the previous study
* Are willing to participate in the study as an outpatient, make visits to the study center for follow-up evaluation, and agree to comply with all study requirements.

Exclusion Criteria:

* None. All subjects who meet the inclusion criteria above may participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of subjects who have been treated with imiquimod or with placebo in one of the aformentioned studies and who demonstrated complete clearance of all clinically visible or palpable AK lesions in the selected treatment area at the end-of-study visit.
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2008-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Levy, MD, Study Director — Graceway Pharmaceuticals, LLC

REFERENCES:
- [Derived] Hanke CW, Swanson N, Bruce S, Berman B, Kulp J, Levy S. Complete clearance is sustained for at least 12 months after treatment of actinic keratoses of the face or balding scalp via daily dosing with imiquimod 3.75% or 2.5% cream. J Drugs Dermatol. 2011 Feb;10(2):165-70. PMID 21283921

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 3b longitudinal and observational study.
Pre-assignment Details: Subjects previously enrolled in studies GW01-0702, GW01-0703, GW01-0704, or GW01-0705 and were completely cleared of their actinic keratosis (AK) lesions in the selected treatment area at the 8-week post-treatment (end-of-study [EOS]) visit returned for follow-up visits at 6 and 12 months after the EOS visit or until a recurrence of AKs.
Groups:
- 2-Week Treatment Group: Subjects who previously enrolled in studies GW01-0702 and GW01-0704 and were completely cleared of their actinic keratosis (AK) lesions in the selected treatment area at the 8-week post-treatment (end-of-study [EOS]) visit returned for follow-up visits at 6 and 12 months after the EOS visit or until a recurrence of AKs.
- 3-Week Treatment Group: Subjects who previously enrolled in studies GW01-0703 and GW01-0705 and were completely cleared of their actinic keratosis (AK) lesions in the selected treatment area at the 8-week post-treatment (end-of-study [EOS]) visit returned for follow-up visits at 6 and 12 months after the EOS visit or until a recurrence of AKs.
Period: Overall Study
Arm/Group | 2-Week Treatment Group | 3-Week Treatment Group
Started | 89 | 90
Completed | 87 | 83
Not Completed | 2 | 7
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2-Week Treatment Group | 3-Week Treatment Group | Total
Number analyzed (Participants) | 89 | 90 | 179
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 50 | 92
  >=65 years | 47 | 40 | 87
Age Continuous [Mean (Standard Deviation); unit: years] | 65.0 (10.9) | 64.0 (10.2) | 64.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 18 | 43
  Male | 64 | 72 | 136
Region of Enrollment [Number; unit: participants]
  United States | 89 | 90 | 179

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrence of AK Lesions
Description: The primary efficacy variable in this study was the absence of AK lesions(sustained clearance rate) in the previously treated area.
Time Frame: Up to one year
Population: Efficacy analyses were conducted on the evaluable subject population defined as all subjects who were eligible and enrolled in the follow-up study. All results were summarized overall and by original Phase 3 randomized treatment regimen and dose group. Actinic keratosis recurrence was categorized by presence or absence only.
Measure: Number; unit: participants
Arm/Group | 2-Week Treatment Group | 3-Week Treatment Group
Number analyzed (Participants) | 89 | 90
participants | 52 | 41

ADVERSE EVENTS:
Time Frame: 12 months
Description: All AEs that were ongoing or started in the previous treatment area at the end of Phase 3 study, or any AEs that occurred that were related to the previous Phase 3 study medication were recorded.
Arm/Group | 2-Week Treatment Group | 3-Week Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/90
Other Adverse Events (participants affected / at risk) | 3/89 | 0/90
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2-Week Treatment Group (N=89) | 3-Week Treatment Group (N=90)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No